CLINICAL TRIAL: NCT00675441
Title: A Phase II Study of Lenalidomide (Revlimid®) as Second Line Therapy in Patients With Chronic Graft-Versus-Host Disease (GVHD)
Brief Title: Lenalidomide (Revlimid®) as Second Line Therapy in Patients With Chronic Graft-Vs-Host Disease (GVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0321
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Graft-versus-Host Disease
Keywords: Chronic Graft-versus-Host Disease; cGVHD; GVHD; Lenalidomide; Revlimid; CC-5013; Stem Cell Transplant; Allogeneic hematopoietic stem cell transplantation; Allogeneic HSCT; HSCT; Post-Transplant Prophylactic Immunosuppressive Therapy; Steroids; Standard-of-care steroid treatment; Corticosteroids; Prednisone; Medrol
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide 10 mg (capsule) by mouth on days 1-21 of a 28-day cycle, for a total of 6 cycles.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg (capsule) by mouth on days 1-21 of a 28-day cycle, for a total of 6 cycles.
  Other Names: Revlimid; CC-5013

SUMMARY:
The goal of this clinical research study is to learn if Revlimid® (lenalidomide), along with standard-of-care steroid treatment you are already receiving, can help to control Chronic Graft-Versus-Host Disease (cGVHD). The safety of this study drug in combination with the steroids will also be studied.

Primary Objectives:

* To assess the response rate of chronic GVHD to Lenalidomide after failing steroids
* To evaluate the safety and tolerability of Lenalidomide in patients with chronic GVHD

Secondary Objectives:

* To assess the steroid-sparing capacity of Lenalidomide (as proportion of patients able to discontinue steroids while receiving or following therapy with Lenalidomide)
* To assess changes in QOL after treatment with Lenalidomide
* To analyze survival at 6 and 12 months after initiation of Lenalidomide
* To evaluate relapse of underlying malignancy as well as second malignancies at 6 and 12 months after initiation of Lenalidomide

DETAILED DESCRIPTION:
The Study Drug:

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. It may decrease or prevent the growth of cancer cells.

Researchers want to find out if lenalidomide can improve the cGVHD and if it can help decrease the amount of steroids you need, which may help prevent long-term side effects that occur when steroids are used over a long period of time.

Study Treatment:

If you are found to be eligible to take part in this study, you will take lenalidomide by mouth (1 larger-dose capsule or 2 smaller-dose capsules) once daily for 21 days followed by 7 days without treatment (a "rest period"). Each 28-day period is called a cycle of therapy. You will have up to 6 cycles of therapy on this study.

Study Drug Administration:

You will swallow lenalidomide capsules whole with water (about 16 ounces) at the same time each day. You should not break, chew, or open capsules. If you miss a dose of lenalidomide, you should take it as soon as you remember on the same day. If you miss taking your dose for the entire day, you will take your regular dose the next day ( DO NOT take double your regular dose to make up for the missed dose).

Study Visits:

During treatment, you will have additional testing to check for side effects and to learn your body's response to therapy. You will have these tests every 2 weeks (during Cycles 1 and 2), once a month (during Cycles 3-6), and every 3 months for up to 1 year from when you started treatment with the study drug.

* You will have a physical exam.
* You will have a full skin assessment. For this assessment, the study doctor will look at your skin to see if your skin shows a reaction to the cGVHD transplant.
* You will have a 2-minute walking test. For this test, you will be asked to walk for 2 minutes, and your walking distance will be measured.
* You will have a grip strength test. For this test, you will be asked to sit down and squeeze something that has a meter to measure your strength.
* You will complete some questionnaires about how you are feeling physically, emotionally, and socially. It should take about 20 minutes to complete.
* You will complete another questionnaire about how you assess your symptoms. It should take about 20 minutes to complete.
* You will have blood drawn (about 2 tablespoons) for routine tests and to check immune-suppressive drug (such as tacrolimus or cyclosporine) levels in your blood.
* You will be asked about how you are feeling and about any side effects you may have experienced since your last visit.

Females who are able to have children that have regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at the end of the study, and 28 days following the end of the study. If your menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following discontinuation from the study.

Your dose of the study drug will be temporarily stopped or decreased if the study doctor thinks it is necessary for your safety. Other drugs may also be given to you to help decrease side effects. The study doctor will tell you what these drugs will be if this is necessary.

Length of Study:

You will be taken off this study if the disease gets worse or you experience any intolerable side effects. If you are tolerating and responding to the study treatment, you will be on this study for up to 1 year from enrollment.

This is an investigational study. Lenalidomide is FDA approved and commercially available for the treatment of specific types of myelodysplastic syndrome (MDS). It is also approved in combination with dexamethasone for previously treated multiple myeloma. Its use in this study is investigational and authorized for use in research only. Up to 46 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic GVHD following allogeneic HSCT of any source (bone marrow, peripheral blood or cord blood stem cells), from any donor type (related, unrelated, mismatched) and with any type of malignancy.
2. Patients must have failed a trial of steroids and calcineurin inhibitors. Steroids must have been given at an initial dose of 1 mg/kg/d of methylprednisolone (MP) or equivalent in combination with tacrolimus or cyclosporine. Steroid refractoriness or resistance will be defined as: 1- Lack of any response after 1 month of treatment with MP, including 15 days of at least 0.5 mg/kg/d, 2- Worsening of existing GVHD or new organ involvement at any time following one week of initiation of MP at 1 mg/kg/day, 3- Reflare or worsening of GVHD at any time during steroid taper.
3. Patients may have received steroids and calcineurin inhibitors (i.e. cyclosporine or tacrolimus) for chronic GVHD. Patients who have previously been treated for chronic GVHD with any other drug or treatment may be enrolled, provided the other drug or treatment was completed >/= 30 days before registration for study entry.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
5. White Blood Count (WBC) >/= 2,500/mm^3, Absolute neutrophil count (ANC)>/= 1,000/mm^3, platelet count >/= 50,000/mm^3
6. Left ventricular ejection fraction >/= 40%. No uncontrolled arrythmias or symptomatic heart disease. forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusion capacity of lung for carbon monoxide (DLCO) >/= 40%.
7. Serum creatinine <2.0 mg/dL. Serum bilirubin <3 * upper limit of normal (ULN), aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transminase (SGOT) and Alanine transaminase (ALT)/ serum glutamic pyruvic transaminase (SGPT) < or = 5 * ULN. No evidence of chronic active hepatitis or cirrhosis.
8. No uncontrolled infections.
9. No evidence of malignancy (patients must be in complete remission from their malignancy)
10. Patients must be able to provide written informed consent, and be 18 years or older at the time of signing consent.
11. Patient must be able to return to clinic for follow up at least every 2 weeks for the first 2 months and at least monthly thereafter.
12. Women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study drug and must either commit to continued abstinence from heterosexual intercourse or agree to use 2 contraceptive methods. These birth control methods must be used for at least 4 weeks before, during and after lenalidomide therapy. Men must agree not to father a child and agrees to use a condom if his partner is of child bearing potential.
13. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. (patients intolerant to ASA may use low molecular weight heparin).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of Lenalidomide.
8. Use of prior immunosuppressants other than steroids and calcineurin inhibitors (i.e. cyclosporine or tacrolimus).
9. Known positive for HIV or infectious hepatitis, type A, B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 04/16/2008 to 12/01/2010. All participants were recruited at The University of Texas MD Anderson Cancer Center medical clinics.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 5
Completed | 2
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
Age Continuous [Median (Full Range); unit: years] | 55 [35 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants' With Treatment Response of Complete or Partial Response
Description: Treatment responses defined as complete (CR) or partial organ response (PR) of chronic Graft-Versus-Host Disease (GVHD) to lenalidomide. Complete organ response (CR) indicates resolution of all reversible manifestations related to chronic GVHD in a specific organ. Partial organ response (PR) requires at least 50% improvement in scale used to measure disease manifestations related to chronic GVHD. Tools for response evaluation were skin assessment and functional assessment including minute walk and grip strength.
Time Frame: Response assessed after completing 28 day cycle, repeated with each cycle for 6 cycles, approximately 180 days.
Population: Of the five (5) participants enrolled, two participants were taken off study after only a few days of therapy and one participant expired, all three of which were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=5)
Sudden Cardiac Arrest (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
The study did not meet all primary and secondary objectives due to slow patient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No